CLINICAL TRIAL: NCT02419794
Title: Recovery by Endovascular Salvage for Cerebral Ultra-acute Embolism (RESCUE)-Japan Registry 2
Status: Completed | Type: Observational
Sponsor: Hyogo Medical University (Other)
Responsible Party: Principal Investigator, Shinichi Yoshimura, Professor, Hyogo Medical University
Other Study IDs: UMIN000015273
Record Dates: First submitted 2015-01-19; First posted 2015-04-17 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group with endovascular treatment: Group with additional endovascular treatment
  Interventions: Procedure: endovascular treatment
- Group without endovascular treatment: Group without additional endovascular treatment

INTERVENTIONS:
Procedure: endovascular treatment — endovascular treatment for acute ischemic stroke patients with large vessel occlusion
  Groups: Group with endovascular treatment

SUMMARY:
The aim of this study is to clarify treatment status and clinical results of acute cerebral ischemia after approval of clot retriever in Japan, and also to obtain a basis for comparative studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted from Oct. 1st 2014 to Sep. 30st 2016.
* Patients who were 20 years and older admitted within 24 hours after onset.
* The patients with large vessel occlusion (ICA, MCA, VA, BA, PCA).
* Patients who did not fulfill the criteria of RESCUE-Japan RCT.

Exclusion Criteria:

･Patients who are considered inappropriate to participate in the study are excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute cerebral large vessel occlusion admitted within 24 hours after onset.
Sampling Method: Non-Probability Sample
Enrollment: 2420 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) of 0-2 at 90 days (+/- 10 days) after onset | 90 days

SECONDARY OUTCOMES:
Death within 90 days (+/- 10 day) after the onset | 90 days
modified Rankin Scale (mRS) of 0-1 at 90 days (+/- 10 days) after onset | 90 days
All bleeding within 90 days (+/- 10 days) after onset | 90 days
All intracranial hemorrhage within 90 days (+/- 10 days) after onset | 90 days
Symptomatic intracranial hemorrhage within 90 days (+/- 10 days) after onset | 90 days

OTHER OUTCOMES:
Symptomatic intracranial hemorrhage within 72 hours (+/- 8 hours) after onset | 72 hours
Reccurrence of stroke within 90 days (+/- 10 days) after onset | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Shinichi Yoshimura, MD, PhD, Principal Investigator — Hyogo Medical University
Locations (1):
- Hyogo College of Medicine, Nishinomiya, Hyōgo, Japan

REFERENCES:
- [Derived] Kamogawa N, Tanaka K, Yamagami H, Yoshimoto T, Uchida K, Morimoto T, Imamura H, Sakai N, Ohara N, Matsumoto Y, Takeuchi M, Shigeta K, Toyoda K, Yoshimura S. Outcomes of Symptomatic Anterior Large Vessel Occlusion by Initial Imaging Assessment Using Diffusion-Weighted Imaging Versus Noncontrast Computed Tomography. Stroke Vasc Interv Neurol. 2022 Apr 16;2(5):e000170. doi: 10.1161/SVIN.121.000170. eCollection 2022 Sep. PMID 41584006
- [Derived] Tanaka K, Yamagami H, Yoshimoto T, Uchida K, Morimoto T, Toyoda K, Sakai N, Yoshimura S. Endovascular Therapy for Acute Ischemic Stroke in Patients With Prestroke Disability. J Am Heart Assoc. 2021 Aug 3;10(15):e020783. doi: 10.1161/JAHA.121.020783. Epub 2021 Jul 21. PMID 34284599
- [Derived] Fujita K, Tanaka K, Yamagami H, Yoshimoto T, Uchida K, Morimoto T, Imamura H, Sakai N, Ohara N, Matsumoto Y, Takeuchi M, Shigeta K, Toyoda K, Yoshimura S. Outcomes of Large Vessel Occlusion Stroke in Patients Aged >/=90 Years. Stroke. 2021 May;52(5):1561-1569. doi: 10.1161/STROKEAHA.120.031386. Epub 2021 Mar 1. PMID 33641385
- [Derived] Saito T, Itabashi R, Yazawa Y, Uchida K, Yamagami H, Sakai N, Morimoto T, Yoshimura S; RESCUE-Japan Registry 2 Investigators. Clinical Outcome of Patients With Large Vessel Occlusion and Low National Institutes of Health Stroke Scale Scores: Subanalysis of the RESCUE-Japan Registry 2. Stroke. 2020 May;51(5):1458-1463. doi: 10.1161/STROKEAHA.119.028562. Epub 2020 Apr 16. PMID 32295504
- [Derived] Yoshimura S, Sakai N, Uchida K, Yamagami H, Ezura M, Okada Y, Kitagawa K, Kimura K, Sasaki M, Tanahashi N, Toyoda K, Furui E, Matsumaru Y, Minematsu K, Morimoto T. Endovascular Therapy in Ischemic Stroke With Acute Large-Vessel Occlusion: Recovery by Endovascular Salvage for Cerebral Ultra-Acute Embolism Japan Registry 2. J Am Heart Assoc. 2018 Apr 25;7(9):e008796. doi: 10.1161/JAHA.118.008796. PMID 29695384